CLINICAL TRIAL: NCT06410794
Title: Work-related Attention Bias Modification Training and Virtual Reality Training in Occupational Rehabilitation: A Multisite Pilot Study
Brief Title: Virtual Reality Training in Occupational Rehabilitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Molde University College (Other)
Collaborators: Norwegian National Advisory Unit on Occupational Rehabilitation (Unknown)
Responsible Party: Principal Investigator, Anita Dyb Linge, Research and Developement Manager, Molde University College
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 254368
Record Dates: First submitted 2024-04-23; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Musculoskeletal Diseases; Mental Health Disorder; Back Pain, Low; Anxiety Disorders; Depression
Keywords: Virtual reality; gaming; occupational rehabilitation; patient experience; quanitative study; qualitative study
MeSH Terms: conditions — Musculoskeletal Diseases; Mental Disorders; Low Back Pain; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This is a non-randomised controlled experiment where we aim to recruit 20 patients from each of the six clinics involved in ABM training and up 100 from each of the clinics involved in VR. That is, 10 receiving ABM training and 10 in the control group, and 60 receiving VR and 40 in the control group. The participants will complete the questionnaires and cognitive measures one the day of arrival and on the penultimate or ultimate day of the rehabilitation/treatment. The measures will take approximately one hour to complete at each measurement point and will not interfere with the participation in the rehabilitation/treatment.
  In the qualitative part of this pilot, it is aimed to recruit 15 patients, five at each of the three clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparing VR training and ABM training (Experimental): The objective of this study is to investigate whether VR and ABM training increases work ability, work-related self-efficacy, attention and reduces symptoms of depression and anxiety and consequently change an attentional bias from negative to positive stimuli. We will compare patients receiving work-related interventions + VR, work-related interventions + ABM training and work-related interventions only. We will also investigate whether positive changes in attentional bias are associated with increased work participation. Self-reported work ability, self-efficacy, depression, anxiety and objective computerised cognitive and emotional testing will be assessed at baseline (start rehabilitation/treatment) and at posttest (end rehabilitation/treatment).
  Interventions: Device: Virtual Reality with Beat Saber
- Patients' experiences with the usage of VR. (No Intervention): The objective of this part is to investigate the experiences in using VR. R&D personell will make individual interviews with five patients at each of the three clinics involved in piloting VR. The aim of the interviews will be to capture how the patients experienced the VR activity, the demands of the VR activity, how VR has influenced different aspects of health and whether VR has influenced the abilities to return to work.

INTERVENTIONS:
Device: Virtual Reality with Beat Saber — The VR activity used in the intervention was an add-on activity that did not replace any other activities in the programme. The off-the-shelf product Beat Saber (Beat Games, Prague, The Czech Republic) is the VR game of choice in our study. In collaboration with the participating clinics a systematic VR activity plan will be developed. This includes the selection of games and designing a plan that is interesting and motivating both for patients and clinicians.
  Arms: Comparing VR training and ABM training

SUMMARY:
Work-related attention bias modification training and virtual reality training in occupational rehabilitation is a multisite pilot study.

The quantitative aim of this pilot study is to compared virtual reality (VR) training and attention bias modication (ABM) training to investigate whether the different training forms result in different results measured with work-related outcomes and cognitive outcomes. The qualitative aim of this pilot study is to investigate the patients' experiences with the usage of VR.

Three rehabilitation insitutions will be recruiting patients participating in occupational rehabilitation, and the study will compare the outcomes of work-related interventions with and without the addition of ABM or VR training.

The study seeks to determine if these interventions can improve work ability, reduce symptoms of depression and anxiety, and change attentional bias from negative to positive stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 67 years
* Must be on sick leave, work assessment allowance or on disability pension
* Receiving work-related rehabilitation or treatment at clinics with either an International Classification of Primary Care, Second edition (ICPC-2) within the musculoskeletal (L), psychiatric (P) or unspecific disorders (A) categories or International Classification Disorders-10 diagnosis within the mental and behavioral disorders (F), Diseases of the musculoskeletal system and connective tissue (M) or other diagnoses.

Exclusion Criteria:

* Applying for a full disability pension;
* Unable to complete the measures and receive instructions in Norwegian.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Increase work ability | Baseline and discharge (four weeks), and 6 and 12 months after discharge
  Self-reported questionnaire measures, (Work Ability Scale). Work ability: Self-rated work ability was assessed using a single-item question to determine the WAS; this question was published by Gould et al. as part of the full work ability index (WAI). The question used by this study to measure WAS ("current work ability compared with your lifetime best") used a scale of 0 to 10 (0 = "completely unable to work" and 10 = "work ability at its best"). The following measurement classification from Gould et al. [46] was used: poor (0 to 5), moderate (6 to 7), good (8 to 9) and excellent (10).
Reduced depression and anxiety | Baseline and discharge (four weeks)
  Self-reported questionnaire measure, (The Hospital Anxiety And Depression Scale).
Increase expectations to return to work | Baseline and discharge (four weeks), and 6 and 12 months after discharge
  Self-reported questionnaire measures, (Return-to-Work Expectation)

SECONDARY OUTCOMES:
Increased cognitive performance and attention | Baseline and discharge (four weeks)
  Computerized cognitive measures.
  - Rapid Visual Information Processing (Cambridge Cognition, 2020). The mean response latency on trials where the subject responded correctly. Calculated across all assessed trials.
Increased cognitive performance and memory | Baseline and discharge (four weeks)
  Computerized cognitive measures.
  - Spatial Working Memory (Cambridge Cognition, 2020). The number of times the subject incorrectly revisits a box in which a token has previously been found.
Increased cognitive performance | Baseline and discharge (four weeks)
  Computerized cognitive measures.
  - Stop Signal Task (Cambridge Cognition, 2020). The estimate of time when an individual can successfully inhibit their responses 50% of the time.
Patients's experiences in using VR | From discharge up to 5 month after discharge.
  Interview guide based on the participants experience.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Jensen, PhD, Study Director — Norwegian National Advisory Unit on Occupational Rehabilitation
Locations (1):
- Norwegian National Advisory Unit on Occupational Rehabilitation, Rauland, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT06410794/Prot_ICF_000.pdf